CLINICAL TRIAL: NCT01560923
Title: A Randomized, Double-Blind Phase II Study of Sipuleucel-T (Provenge®) Followed by Indoximod or Placebo in the Treatment of Patients With Asymptomatic or Minimally Symptomatic Metastatic Castration Resistant Prostate Cancer
Brief Title: Phase II Study of Sipuleucel-T and Indoximod for Patients With Refractory Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011LS109
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Results first posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Metastatic Prostate Cancer
Keywords: hormone refractory prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 1-methyltryptophan; sipuleucel-T

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sipuleucel-T + Oral Indoximod (Experimental): Oral Indoximod will be self-administered by mouth twice daily (1200 mg) for 6 months starting after the last (3rd) infusion of sipuleucel-T. Indoximod is a sterile tan powder compounded in capsule form of 200 mg.
  Interventions: Biological: Indoximod; Biological: Sipuleucel-T
- Sipuleucel-T + Placebo (Placebo Comparator): Placebo is identical-looking to Indoximod and provided in the same manner.
  Interventions: Biological: Sipuleucel-T; Other: Placebo

INTERVENTIONS:
Biological: Indoximod — Given twice daily (1200 mg total) by mouth for 6 months.
  Other Names: 1-methyl-D-tryptophan
  Arms: Sipuleucel-T + Oral Indoximod
Biological: Sipuleucel-T — Sipuleucel-T will be administered as standard of care. Given by infusion over 60 minutes at Week 0, 2 and 4. Patients will undergo leukapheresis at weeks 0, 2, and 4 with sipuleucel-T infused 3 days later (i.e. Monday/Thursday; Tuesday/Friday).
  Other Names: Provenge
Other: Placebo — Given in same manner as Indoximod; 1200 mg per day by mouth.
  Arms: Sipuleucel-T + Placebo

SUMMARY:
This is a randomized, double blind, multi-institutional phase II therapeutic study of Indoximod or placebo after the completion of standard of care sipuleucel-T (Provenge®) in men with asymptomatic or minimally symptomatic metastatic prostate cancer that is castration resistant (hormone refractory). Patients are randomized to receive either twice daily oral Indoximod or placebo for 6 months beginning the day after the third and final sipuleucel-T infusion.

DETAILED DESCRIPTION:
Sipuleucel-T will be administered as standard of care. Oral Indoximod/placebo will be self-administered twice daily for 6 months starting after the last infusion of sipuleucel-T. Patients will be treated for a minimum of 12 weeks of Indoximod/placebo before disease progression can be declared and Indoximod/placebo will not be discontinued for increasing prostate specific antigen (PSA) in the absence of symptomatic clinical progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented adenocarcinoma of the prostate with metastatic disease as evidenced by soft tissue and/or bony metastases on baseline computed tomography (CT) scan of the abdomen and pelvis and/or bone scan
* Castration-resistant based on a current or historical evidence of disease progression despite surgical or medical castration as demonstrated by one or more of the following:

  * PSA progression (defined as two consecutive prostate specific antigen (PSA) measurements at least 14 days apart ≥ 2.0 ng/ml and ≥ 50% above the minimum PSA during castration therapy or above pre-treatment value if no response)
  * progression of measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) criteria (≥ 50% increase in the sum of the cross products of all measurable lesions or the development of any new lesions
  * progression of non-measureable disease
* Serum PSA ≥ 2.0 ng/ml at study enrollment
* Castration levels of testosterone defined as ≤ 30 ng/dL at study enrollment. Must be at least 3 months from surgical castration or must have received medical castration therapy for at least 3 months and be receiving such therapy at the time of confirmed disease progression
* Asymptomatic or minimally symptomatic disease as demonstrated by Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1 and no need for opiate pain medications to control pain/symptoms
* Age 18 years and old
* Adequate bone marrow, renal and hepatic function within 14 days of study enrollment defined as:

  * Bone marrow: WBC > 3,000/uL; absolute neutrophil count > 1,500/uL; platelets > 100,000/uL
  * Renal: creatinine within institutional upper limit of normal (ULN) OR creatinine clearance > 60 mL/min/1.73 m2 for patients with creatinine levels above ULN
  * Hepatic: total bilirubin < 1.5 X institutional ULN; aspartate aminotransferase (AST ((SGOT)) and alanine aminotransferase (ALT((SGPT)) < 2.5 X institutional ULN

Exclusion Criteria:

* Chronic steroid dependence (should stop all steroid supplementation 4 weeks prior to enrollment)
* Human immunodeficiency virus (HIV)-positive patients and those with other acquired/inherited immunodeficiency
* History of gastrointestinal disease causing malabsorption or obstruction such as, but not limited to Crohn's disease, celiac sprue, tropical sprue, bacterial overgrowth/blind loop syndrome, gastric bypass surgery, strictures, adhesions, achalasia, bowel obstruction, or extensive small bowel resection
* Inability to take medications by mouth
* History of allergic reactions attributed to compounds of similar chemical or biologic composition
* Active autoimmune disease, chronic inflammatory condition, conditions requiring concurrent use of any systemic immunosuppressants or steroids. Mild-intermittent asthma requiring only occasional beta-agonist inhaler use or mild localized eczema will not be excluded.
* Previous allo-transplant of any kind
* History of prior treatment with anti-CTLA4 blocking antibody

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shilpa Gupta, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (4):
- United States (4):
  - University of Illinois Medical Center, Chicago, Illinois
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - New York Presbyterian/Weill Cornell Medical Center, New York, New York
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient withdrew or refused to participate after receiving protocol therapy
Period: Overall Study
Arm/Group | Sipuleucel-T + Placebo | Sipuleucel-T + Oral Indoximod
Started | 24 | 22
Completed | 24 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control (Placebo) Arm: Placebo is identical-looking to Indoximod and provided in the same manner.
  Sipuleucel-T: Sipuleucel-T will be administered as standard of care. Given by infusion over 60 minutes at Week 0, 2 and 4. Patients will undergo leukapheresis at weeks 0, 2, and 4 with sipuleucel-T infused 3 days later (i.e. Monday/Thursday; Tuesday/Friday).
  Placebo: Given in same manner as Indoximod; 1200 mg per day by mouth.
- Treatment: Oral Indoximod will be self-administered by mouth twice daily (1200 mg) for 6 months starting after the last (3rd) infusion of sipuleucel-T. Indoximod is a sterile tan powder compounded in capsule form of 200 mg.
  Indoximod: Given twice daily (1200 mg total) by mouth for 6 months.
  Sipuleucel-T: Sipuleucel-T will be administered as standard of care. Given by infusion over 60 minutes at Week 0, 2 and 4. Patients will undergo leukapheresis at weeks 0, 2, and 4 with sipuleucel-T infused 3 days later (i.e. Monday/Thursday; Tuesday/Friday).
- Total: Total of all reporting groups
Arm/Group | Control (Placebo) Arm | Treatment | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 9 | 15
  >=65 years | 18 | 13 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 24 | 22 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 22 | 22 | 44
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 23 | 16 | 39
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Immune Response to Sipuleucel-T
Description: Assess the augmentation of immune response (PA2024) to sipuleucel-T measured at 14 weeks from first leukapheresis, in response to twice daily oral Indoximod at a dose of 1200 mg/day or an identical looking placebo.
  The frequency of antigen specific, cytokine producing cells will be determined by an ELISPOT assay. ELISPOT assay will use whole PBMC to assess interferon gamma production in response to the immunizing protein PA2024. Increase in number of ELISPOT responses to PBMC in patients in the treatment arm will be compared to those in control arm.
Time Frame: 14 Weeks from First Leukapheresis
Measure: Geometric Mean (95% Confidence Interval); unit: Spots per ml
Arm/Group | Sipuleucel-T + Placebo | Sipuleucel-T + Oral Indoximod
Number analyzed (Participants) | 24 | 22
Spots per ml | 29.6 [4.86 to 180.37] | 25.45 [2.92 to 222.12]

2. Secondary Outcome: Number of Participants With Progression Free Survival at 6 Months
Description: Progression free survival (PFS) is a composite endpoint defined as disease progression in bone or soft tissues, PSA progression, worsening pain, or death. PFS will be measured in months from the time of study enrollment until the date of disease progression.
  Progression is evaluated using the international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) [Eur J Ca 45:228-247, 2009]. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Sipuleucel-T + Placebo | Sipuleucel-T + Oral Indoximod
Number analyzed (Participants) | 24 | 22
Participants | 6 | 11

3. Secondary Outcome: Objective Response Rate
Description: rate as defined by Prostate Cancer Working Group -2 (PCWG2). ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST)(version 1.1) Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesion.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sipuleucel-T + Placebo | Sipuleucel-T + Oral Indoximod
Number analyzed (Participants) | 24 | 22
Participants
  Partial response (PR) | 1 | 0
  Not Evaluable | 0 | 2
  Stable Disease (SD) | 5 | 11
  Baseline | 3 | 1
  Non-CR/Non-PD | 1 | 1
  Progressive Disease (PD) | 12 | 7
  Not Assessed | 2 | 0

4. Secondary Outcome: Overall Survival
Description: To evaluate 2 year overall survival
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Sipuleucel-T + Placebo | Sipuleucel-T + Oral Indoximod
Number analyzed (Participants) | 24 | 22
Participants | 18 | 17

5. Secondary Outcome: Quality of Life Scale Results
Description: measured by the performance status with scale of 0-5 0 being 'normal activity' and 5 'being dead'
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Sipuleucel-T + Placebo | Sipuleucel-T + Oral Indoximod
Number analyzed (Participants) | 24 | 22
Participants
  Baseline Performance Status Score: 0 - Normal activity, Fully active | 19 | 15
  Baseline Performance Status Score: 1- Symptoms but ambulatory | 5 | 7
  Baseline Performance Status Score: No Data | 0 | 0
  Post Treatment performance Status Score: 0 - Normal activity, Fully active | 7 | 9
  Post Treatment performance Status Score: 1- Symptoms but ambulatory | 10 | 3
  Post Treatment performance Status Score: No Data | 7 | 10

6. Secondary Outcome: Ratio of Antibodies to PA2024
Description: Assess the augmentation of immune response (PA2024) to sipuleucel-T measured at 14 weeks from first leukapheresis, in response to twice daily oral Indoximod at a dose of 1200 mg/day or an identical looking placebo.
  The frequency of antigen specific, cytokine producing cells will be determined by an ELISPOT assay. ELISPOT assay will use whole PBMC to assess interferon gamma production in response to the immunizing protein PA2024.
  Antibodies to PA2024 is measured by ELISA. The ratio of antibodies to ELISPOT responses to PBMC in patients in the treatment arm will be compared to those in control arm.
Time Frame: 14 Weeks from First Leukapheresis
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Sipuleucel-T + Placebo | Sipuleucel-T + Oral Indoximod
Number analyzed (Participants) | 24 | 22
Ratio
  PA2024 IGG ratio (wk14/baseline) | 13.05 [5.05 to 33.72] | 9.19 [3.04 to 27.8]
  PA2024 IGGIGM ratio (wk14/baseline) | 104.39 [33.88 to 321.66] | 111.43 [35.49 to 349.89]

ADVERSE EVENTS:
Time Frame: 28 days
Groups:
- Sipuleucel-T + Indoximod: Oral Indoximod will be self-administered by mouth twice daily (1200 mg) for 6 months starting after the last (3rd) infusion of sipuleucel-T. Indoximod is a sterile tan powder compounded in capsule form of 200 mg.
  Indoximod: Given twice daily (1200 mg total) by mouth for 6 months.
  Sipuleucel-T: Sipuleucel-T will be administered as standard of care. Given by infusion over 60 minutes at Week 0, 2 and 4. Patients will undergo leukapheresis at weeks 0, 2, and 4 with sipuleucel-T infused 3 days later (i.e. Monday/Thursday; Tuesday/Friday).
Arm/Group | Sipuleucel-T + Indoximod | Sipuleucel-T + Placebo
All-Cause Mortality (participants affected / at risk) | 5/22 | 6/24
Serious Adverse Events (participants affected / at risk) | 2/22 | 1/24
Other Adverse Events (participants affected / at risk) | 20/22 | 21/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sipuleucel-T + Indoximod (N=22) | Sipuleucel-T + Placebo (N=24)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sipuleucel-T + Indoximod (N=22) | Sipuleucel-T + Placebo (N=24)
Positive ANA panel 1:320 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymph node pain (bilateral inguinal) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
White blood cell count decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 2 (2)
Watering eyes (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 0 (0)
Bloating (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (6) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 6 (10)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Increased appetite (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 4 (5)
Mouth sores (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal Mucus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (2) | 1 (1)
Teeth discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
GERD (Gastrointestinal disorders) | 1 (3) | 2 (2)
Chills (General disorders) | 1 (1) | 3 (4)
TMJ pain (General disorders) | 0 (0) | 1 (1)
Fatique (General disorders) | 9 (11) | 7 (10)
Fever (General disorders) | 3 (3) | 2 (2)
Flu like symptoms (General disorders) | 1 (1) | 3 (3)
Other general disorders -Reflux (General disorders) | 0 (0) | 2 (3)
Pain (General disorders) | 1 (1) | 5 (13)
Edema (General disorders) | 2 (2) | 2 (2)
Chest pressure (General disorders) | 0 (0) | 1 (1)
Toe fungal infection (Infections and infestations) | 1 (2) | 0 (0)
Toxoplasma exposure (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2) | 1 (1)
right leg infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (2)
Papular rash to nose and left neck (Infections and infestations) | 1 (1) | 0 (0)
Left fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Issues with return IV (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bleeding to cather (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Elevated alkaline phosphatase (Investigations) | 1 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Anemia (Investigations) | 1 (1) | 0 (0)
Weight gain (Investigations) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia, intermittent (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (8) | 7 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 4 (4)
Memory loss (Nervous system disorders) | 2 (2) | 0 (0)
Nueropathy (Nervous system disorders) | 0 (0) | 2 (2)
Paresthesia (Nervous system disorders) | 1 (1) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary hesitancy (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder incontinence (Renal and urinary disorders) | 0 (0) | 2 (3)
Pelvic pain (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Erectile Dysfunction (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hematuria (Vascular disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 3 (3) | 5 (5)
Hypertension (Vascular disorders) | 3 (3) | 1 (6)
Thromoembolic event (Vascular disorders) | 1 (2) | 0 (0)
Other; Tongue Swelling (General disorders) | 1 (1) | 0 (0)
Other; Spinal tenderness (General disorders) | 1 (1) | 0 (0)
Other; Stiffness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Other; Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Other; Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Other; Slight rash (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0)
Other; Dermatitis Scrotum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Other; Slight thickening of the skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 1 (2) | 1 (1)
Other; Fatigue (General disorders) | 1 (1) | 0 (0)
ecchymois bilateral arms from leukapheresis access site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT01560923/Prot_SAP_000.pdf